CLINICAL TRIAL: NCT05402267
Title: The Effects of Exosomes in Children With Adenoid Hypertrophy Accompanied by Otitis Media With Effusion
Brief Title: The Effects of Exosomes in Otitis Media With Effusion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: OME-2022
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Otitis Media With Effusion; Adenoid Hypertrophy
MeSH Terms: conditions — Otitis Media with Effusion | interventions — Adenoidectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- OA: OME-Adenoid group: Patients who meet the follow inclusion criteria will be considered eligible as the OME-Adenoid (OA) group
  Interventions: Procedure: Adenoidectomy
- CA: Control-Adenoid group: Patients who meet the follow inclusion criteria will be considered eligible as the Control-Adenoid (CA) group
  Interventions: Procedure: Adenoidectomy
- CO: Control-OME group: Patients who meet the follow inclusion criteria will be considered eligible as the Control-OME (CO) group
- control group: Patients without OME and adenoid hypertrophy will be considered eligible as the control group

INTERVENTIONS:
Procedure: Adenoidectomy — Adenoidectomy will be conducted in OA and CA groups
  Groups: CA: Control-Adenoid group; OA: OME-Adenoid group

SUMMARY:
The particularity of adenoids, as a reservoir of bacterial pathogens and immune molecules, is known to be significantly involved in children with otitis media with effusion (OME). As an important carrier of intercellular substance transfer and signal transduction, exosomes with different biological functions can be secreted by different types of cells. There remains significant uncertainty regarding the clinical transmitter of exosomes to OME, especially in its pathophysiologic development. In this study, the investigators try to elucidate the biological functions of exosomes in children with adenoid hypertrophy accompanied by OME.

Patients with adenoid hypertrophy or otitis media will be separated into three groups: those with adenoid hypertrophy, with otitis media and with adenoid hypertrophy and otitis media both, as well as a healthy control group. Participants in the four groups will have their middle ear effusion, nasopharyngeal secretion, and peripheral blood samples taken, from which exosomes will be separated for further analysis. Adenoidectomy will be conducted in adenoid hypertrophy accompanied by OME and adenoid hypertrophy alone and their adenoid tissue will be collected. Blood will be collected again 3 months after surgery and middle ear and nasopharyngeal examinations will be performed. Exosomes will be isolated for follow-up studies as before surgery. Investigators will also use proteome research, exosome biomarkers, and high-throughput sequencing to examine the pathophysiology of OME, particularly inflammation-related etiology, in order to provide novel ideas for OME diagnosis and treatment.

DETAILED DESCRIPTION:
This study will explore the pathogenesis of OME by detecting the exosome in middle ear fluid, nasopharyngeal secretions and peripheral blood in order to identify areas of opportunity for future research and to provide a theoretical basis for drug development for the treatment of secretory otitis media.

240 subjects will be recruited from Eye and ENT hospital of Fudan University or the community. They will be divided into four groups: adenoid hypertrophy accompanied by OME (group OA, n=60), adenoid hypertrophy alone (group CA, n=60), OME alone (group CO, n=60) and healthy control group (children without OME or adenoid hypertrophy, n=60). All participants will undergo the examinations of middle ear and nasopharynx in addition to blood collection when they get into the groups. The exosomes will be isolated form middle ear effusions, nasopharyngeal secretions/adenoid tissue, and peripheral blood collected from all participants. The OA and CA groups will undergo adenoidectomy and their adenoid tissue will be collected. Blood will be collected again 3 months after surgery and middle ear and nasopharyngeal examinations will be performed. Exosomes will be isolated for follow-up studies as before surgery.

The primary outcome measures will be (1) ANOVA of the alterations and related gene expression of exosome contents in nasopharyngeal secretions in the four groups; (2) microbial alterations and the exosomes from biofilm on the surface of the adenoids in OA and CA groups preoperative and postoperative; and (3) the differences of exosomes from peripheral blood samples in OA and CA groups preoperative and postoperative.

ELIGIBILITY:
Inclusion Criteria:

OME-Adenoid (OA) group:

1. Children aged between 4 and 10 years old.
2. Diagnosis of chronic otitis media with effusion, and the course of disease is at least 3 months.
3. There are varying degrees of hearing loss. PTA (The mean hearing threshold of 500Hz, 1000Hz and 2000Hz) ≥ 30dB.
4. Nasopharyngeal lateral X-ray showing A/N > 0.6 of adenoids.

Control-Adenoid (CA) group:

1. Children aged between 4 and 10 years old.
2. Nasopharyngeal lateral X-ray showing A/N > 0.6 of adenoids.

Control-OME (CO) group:

1. Children aged between 4 and 10 years old.
2. Diagnosis of chronic otitis media with effusion, and the course of disease is at least 3 months.
3. There are varying degrees of hearing loss. PTA (The mean hearing threshold of 500Hz, 1000Hz and 2000Hz) ≥ 30dB.

Exclusion Criteria:

1. Patients who have had one or more episodes of otitis media in the previous one year.
2. Any immunologic diseases.
3. Any intrinsic diseases of hearing system, anatomic or physiologic defect of the ear.
4. Pharmacologic abnormality.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 240 subjects will be recruited from Eye and ENT hospital of Fudan University or the community.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
differential gene expression | 3 months
  ANOVA of the alterations and related gene expression of exosome contents in nasopharyngeal secretions in the four groups
detection of adenoids | 3 months
  microbial alterations and the exosomes from biofilm on the surface of the adenoids in OA and CA groups preoperative and postoperative
detection of exosomes | 3 months
  the differences of exosomes from peripheral blood samples in OA and CA groups preoperative and postoperative

IPD SHARING:
Plan to Share IPD: No